CLINICAL TRIAL: NCT00861003
Title: An Exploratory Study on Comparison of Electronic Monitoring and Other Measures of Adherence to Antipsychotic Medication in Outpatients With Schizophrenia or Schizoaffective Disorder
Brief Title: An Adherence Study of Antipsychotic Medication in Outpatients With Schizophrenia or Schizoaffective Disorder
Acronym: MEMS-SPR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Seung-Hyun Kim, Professor
Other Study IDs: KSH001
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; adherence
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Schizophrenia, antipsychotics: Stable outpatient status of schizophrenia or schizoaffective disorder currently taking a single oral antipsychotic
  Interventions: Device: Medication Event Monitoring System (MEMS)

INTERVENTIONS:
Device: Medication Event Monitoring System (MEMS) — MEMS is a medication vial cap that electronically records the date and time of bottle opening.

SUMMARY:
This prospective study examines the differences among several measures of adherence to antipsychotic medications in outpatients with schizophrenia. Adherence is assessed by using self-report, physician report, pill count and electronic monitoring. The rates of adherence/non-adherence with various tools will be manifested. The association between antipsychotic adherence/non-adherence and various clinical status, including psychotic symptoms, depressive symptoms, side effects, neurocognitive function and insight are analyzed. Participants are assessed at baseline during a visit to their outpatient clinic and followed up for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent
2. Male or female, aged from 20 to 65 years
3. Clinician rendered diagnosis of schizophrenia or schizoaffective disorder documented by a checklist of Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV) criteria
4. Currently taking a single oral antipsychotic (e.g., Quetiapine, Risperidone, Olanzapine, or Amisulpride).
5. Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropine (HCG) test at enrolment
6. Outpatient status, with psychiatric hospitalization or psychiatric emergency room visit within the previous 2 years and no hospitalizations within 3 months
7. mild to moderate symptom checked by CGI-S (less than score 4)
8. Able to understand and comply with the requirements of the study

Exclusion Criteria:

1. Any DSM-IV Axis I disorder not defined in the inclusion criteria
2. Presence of a co-morbid diagnosis that might influence outcome measures (e.g., mental retardation)
3. Alcohol or substance dependence at enrolment (except dependence in full remission, and except for caffeine or nicotine dependence), as defined by DSM-IV criteria
4. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
5. Pregnancy or lactation
6. Evidence of hypersensitivity to Quetiapine or other antipsychotics used in the study
7. Use of any cytochrome P450 inhibitors or inducers in the 14 days preceding enrolment
8. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
9. use of pillbox
10. Treatment with Clozapine (because of its unique monitoring guidelines)
11. Administration of electroconvulsive therapy (ECT) in the last 6 months
12. Unstable or inadequately treated medical condition such as heart, liver, kidney, or lung disease, or a seizure disorder
13. Involvement in the planning and conduct of the other study.
14. Participation in another drug trial within 4 weeks prior enrolment into this study or longer in accordance with local requirements.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinician rendered diagnosis of schizophrenia or schizoaffective disorder documented by a checklist of Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV) criteria
Sampling Method: Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Adherence is assessed by four methods including Medication Event Monitoring System | 8 weeks

SECONDARY OUTCOMES:
Various factors that have been identified as influencing adherence | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea